CLINICAL TRIAL: NCT03414047
Title: A Phase 2 Study of Prexasertib in Platinum-Resistant or Refractory Recurrent Ovarian Cancer
Brief Title: A Study of Prexasertib (LY2606368) in Platinum-Resistant or Refractory Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16712; I4D-MC-JTJN (Other: Eli Lilly and Company); 2017-004009-42 (EudraCT Number)
Record Dates: First submitted 2018-01-12; First posted 2018-01-29 (Actual); Results first posted 2020-06-17 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer
Keywords: DNA damage repair; replication stress
MeSH Terms: conditions — Ovarian Neoplasms | interventions — prexasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Prexasertib Cohort 1 (Experimental): Participants received 105 milligram per square meter (mg/m²) prexasertib as an approximately 60 (+10) minute IV infusion on Day 1 and 15 of a 28-day cycle. Participants were with platinum-resistant disease, breast cancer susceptibility gene (BRCA) negative and have received ≥3 lines of prior therapy.
  Interventions: Drug: Prexasertib
- Prexasertib Cohort 2 (Experimental): Participants received 105 mg/m² prexasertib as an approximately 60 (+10) minute IV infusion on Day 1 and 15 of a 28-day cycle. Participants were with platinum-resistant disease, BRCA negative and have received <3 lines of prior therapy.
  Interventions: Drug: Prexasertib
- Prexasertib Cohort 3 (Experimental): Participants received 105 mg/m² prexasertib as an approximately 60 (+10) minute IV infusion on Day 1 and 15 of a 28-day cycle. Participants were with platinum-resistant disease, BRCA positive and received a prior poly ADP ribose polymerase (PARP) inhibitor.
  Interventions: Drug: Prexasertib
- Prexasertib Cohort 4 (Experimental): Participants received 105 mg/m² prexasertib as an approximately 60 (+10) minute IV infusion on Day 1 and 15 of a 28-day cycle. Participants were with platinum refractory disease, BRCA positive or negative, no restriction on number of lines of prior therapy.
  Interventions: Drug: Prexasertib

INTERVENTIONS:
Drug: Prexasertib — Administered IV
  Other Names: LY2606368

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of prexasertib in women with platinum-resistant or refractory recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women who have high-grade serous ovarian, primary peritoneal or fallopian tube cancer.
* Cohorts 1 to 3: Have platinum-resistant disease and have documented test results assessing alterations in the BRCA1 and BRCA2 genes prior to receiving study treatment.
* Cohort 1: Are BRCA negative and have received 3 or more prior lines of therapy.
* Cohort 2: Are BRCA negative and have received less than 3 prior lines of therapy.
* Cohort 3: Are BRCA positive and have previously received a PARP.
* Cohort 4: Have primary platinum refractory disease.
* Have adequate organ function.
* Must be able and willing to undergo mandatory tumor biopsy.

Exclusion Criteria:

* Cohorts 1-3: Have previously received all of the following agents at any time in the platinum-resistant setting: gemcitabine, pegylated liposomal doxorubicin, and paclitaxel.
* Have known central nervous system malignancy or metastasis.
* Have previously participated in any study involving a checkpoint kinase 1 inhibitor or have hypersensitivity to the study drug or excipients.
* Have at least one of the following:

  * history of abdominal fistula or gastrointestinal perforation
  * intra-abdominal abscess within last 3 months prior to the first dose of study drug
  * a radiographically confirmed bowel obstruction within 3 months prior to the first dose of study drug
* Have a symptomatic human immunodeficiency virus infection or symptomatic activated/reactivated hepatitis A, B, or C (screening is not required).
* Have a serious cardiac condition.
* Have a history of prior radiotherapy to the whole pelvis.
* Have chronic daily treatment with corticosteroids, excluding inhaled or topical steroids.
* Have known factors that may increase the risk of infection while on study drug treatment. These may include, but are not limited to, an indwelling peritoneal catheter or open wounds. Catheters for vascular access are permitted.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2020-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (46):
- United States (14):
  - Arizona Oncology Associates, P.C., Tucson, Arizona
  - Kaiser Permanente Medical Center, Vallejo, California
  - University of Southern Florida School of Medicine, Gainesville, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Research Medical Center, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Care Associates, Tulsa, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Sioux Valley Clinic, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Mater Adult Hospital Brisbane, South Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Burnside War Memorial Hospital, Toorak Gardens, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - GZA St Augustinus, Wilrijk
- Israel (3):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Italy (3):
  - Policlinico Univ. Agostino Gemelli, Rome, Lazio
  - Istituto Europeo di Oncologia, Milan, Milan
  - Istituto Tumori Fondazione G. Pascale IRCCS, Napoli, Naples
- South Korea (4):
  - Samsung Medical Center, Seoul, Korea
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- United Kingdom (6):
  - University College Hospital - London, London, Greater London
  - Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Mount Vernon Hospital, Northwood, Middlesex
  - Royal Surrey County Hospital, Guildford, Surrey
  - Royal Marsden Hospital, Sutton, Surrey
  - Northampton General Hospital, Northampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Konstantinopoulos PA, Lee JM, Gao B, Miller R, Lee JY, Colombo N, Vergote I, Credille KM, Young SR, McNeely S, Wang XA, Lin AB, Shapira-Frommer R. A Phase 2 study of prexasertib (LY2606368) in platinum resistant or refractory recurrent ovarian cancer. Gynecol Oncol. 2022 Nov;167(2):213-225. doi: 10.1016/j.ygyno.2022.09.019. Epub 2022 Sep 30. PMID 36192237
- See also: A Study of Prexasertib (LY2606368) in Platinum-Resistant or Refractory Recurrent Ovarian Cancer — https://trials.lillytrialguide.com/en-US/trial/34RLV3dW4MKcsOCsOEICUO

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Completers included participants who died from any cause and participants who were alive and on study (either on study treatment or in long term follow-up) at study conclusion.
Pre-assignment Details: Only 169 participants were assigned to one of the 4 cohorts in this study. Data is not available for 3 participants who discontinued before the start of the treatment.
Period: Overall Study
Arm/Group | Prexasertib Cohort 1 | Prexasertib Cohort 2 | Prexasertib Cohort 3 | Prexasertib Cohort 4
Started | 53 | 46 | 41 | 29
Received at Least One Dose of Study Drug | 53 | 46 | 41 | 29
Completed | 51 | 46 | 38 | 27
Not Completed | 2 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Prexasertib Cohort 1: Participants received 105 mg/m² prexasertib as an approximately 60 (+10) minute IV infusion on Day 1 and 15 of a 28-day cycle. Participants were with platinum-resistant disease, breast cancer susceptibility gene (BRCA) negative and have received ≥3 lines of prior therapy.
- Total: Total of all reporting groups
Arm/Group | Prexasertib Cohort 1 | Prexasertib Cohort 2 | Prexasertib Cohort 3 | Prexasertib Cohort 4 | Total
Number analyzed (Participants) | 53 | 46 | 41 | 29 | 169
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (9.4) | 62.3 (9.4) | 59.5 (8.6) | 59.0 (13.4) | 60.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 46 | 41 | 29 | 169
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 0 | 4
  Not Hispanic or Latino | 48 | 40 | 39 | 28 | 155
  Unknown or Not Reported | 4 | 3 | 2 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 8 | 4 | 3 | 21
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 2
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 46 | 36 | 37 | 25 | 144
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 4 | 5 | 2 | 2 | 13
  Belgium | 4 | 1 | 3 | 0 | 8
  United States | 6 | 13 | 3 | 10 | 32
  United Kingdom | 6 | 9 | 4 | 1 | 20
  Italy | 4 | 4 | 8 | 7 | 23
  Israel | 6 | 3 | 7 | 4 | 20
  Australia | 14 | 7 | 10 | 3 | 34
  Spain | 9 | 4 | 4 | 2 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR): Overall Response Rate (ORR)
Description: Overall response rate is the best response of complete response (CR) or partial response (PR) as classified by the independent central review according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants per cohort with at least 1 measurable lesion, multiplied by 100.
Time Frame: Baseline through Disease Progression (Up to 6 months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Prexasertib Cohort 1 | Prexasertib Cohort 2 | Prexasertib Cohort 3 | Prexasertib Cohort 4
Number analyzed (Participants) | 53 | 46 | 41 | 29
Percentage of Participants | 11.3 [4.3 to 23.0] | 13.0 [4.9 to 26.3] | 12.2 [4.1 to 26.2] | 6.9 [0.8 to 22.8]

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of Prexasertib
Description: Pharmacokinetics(PK): Maximum Plasma Concentration of Prexasertib. The same dose was administered to Cohort 1, 2, 3 and 4 and were combined for analysis.
Time Frame: Cycle 1, Cycle 2, Cycle 4, Cycle 6 (Day 1 (End of prexasertib infusion (+15 min), 1-2 hours following end of prexasertib infusion), Cycle 2, day 1(Prior to start of prexasertib infusion)
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data. Cohort 1, 2, 3 and 4 received the same dose and were combined per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter(ng/mL)
Groups:
- Prexasertib: Participants received 105 mg/m² prexasertib as an approximately 60 (+10) minute IV infusion on Day 1 and 15 of a 28-day cycle. (Participants combined from all the Cohorts 1 to 4)
Arm/Group | Prexasertib
Number analyzed (Participants) | 151
nanograms per milliliter(ng/mL)
  Cycle 1 | 668 (50)
  Cycle 2: number analyzed (Participants) | 105
  Cycle 2 | 718 (62)
  Cycle 4: number analyzed (Participants) | 56
  Cycle 4 | 678 (61)
  Cycle 6: number analyzed (Participants) | 27
  Cycle 6 | 672 (42)

3. Secondary Outcome: Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of CR, PR, or Stable Disease (SD) for at Least 4 Months
Description: DCR is defined as the number of participants who achieve a best overall response of CR, PR or SD for ≥4 months as determined by per RECIST version 1.1. CR is the disappearance of all target and non-target lesions; PR is a ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesion; SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Disease control rate is calculated as a total number of participants with CR or PR or SD divided by the total number of participants treated, then multiplied by 100.
Time Frame: Baseline through Disease Progression (up to 6 months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Prexasertib Cohort 1 | Prexasertib Cohort 2 | Prexasertib Cohort 3 | Prexasertib Cohort 4
Number analyzed (Participants) | 53 | 46 | 41 | 29
Percentage of participants | 45.3 [31.6 to 59.6] | 32.6 [19.5 to 48.0] | 31.7 [18.1 to 48.1] | 31.0 [15.3 to 50.8]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the date measurement criteria for CR or PR (whichever is first recorded) are first met until the first date that disease is recurrent or objective progression is observed, per RECIST 1.1, or the date of death from any cause in the absence of objectively determined disease progression or recurrence. Participants known to be alive and without disease progression will be censored at the time of the last adequate tumor assessment.
Time Frame: Date of CR or PR to Date of Disease Progression or Death Due to Any Cause (up to 20 months)
Population: All randomized participants who received at least one dose of study drug and had CR or PR responses. Number of participants censored Cohort 1 = 0, Cohort 2 = 1, Cohort 3 = 0 and Cohort 4 = 0.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Prexasertib Cohort 1 | Prexasertib Cohort 2 | Prexasertib Cohort 3 | Prexasertib Cohort 4
Number analyzed (Participants) | 6 | 5 | 5 | 2
Months | 8.57 [5.55 to NA] — The upper 95% confidence interval was not achieved due to high censoring rate. | 3.84 [2.79 to NA] — The upper 95% confidence interval was not achieved due to high censoring rate. | 5.55 [3.65 to 9.36] | 5.31 [5.06 to NA] — The upper 95% confidence interval was not achieved due to high censoring rate.

5. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction in CA-125 Levels From Baseline
Description: CA-125 response is defined as ≥50% reduction in CA-125 levels from a pretreatment sample. The response must be confirmed and maintained for ≥28 days according to GCIG criteria. Participants must have a pretreatment sample that is ≥2 times the upper limit of the reference range and obtained within 2 weeks before starting the treatment.
Time Frame: Baseline, 4 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Prexasertib Cohort 1 | Prexasertib Cohort 2 | Prexasertib Cohort 3 | Prexasertib Cohort 4
Number analyzed (Participants) | 53 | 46 | 41 | 29
Percentage of participants | 39.6 | 34.8 | 17.1 | 37.9

6. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival (PFS) is defined as the time from the date of enrollment until the first occurrence of documented disease progression per RECIST 1.1, or death from any cause in the absence of progressive disease (PD). Participants known to be alive and without disease progression will be censored at the time of the last adequate tumor assessment.
Time Frame: Baseline to Disease Progression or Death from any Cause (Up to 22 months)
Population: All randomized participants who received at least one dose of study drug. Number of participants censored Cohort 1 = 6, Cohort 2 = 4, Cohort 3 = 4 and Cohort 4 = 4.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Prexasertib Cohort 1 | Prexasertib Cohort 2 | Prexasertib Cohort 3 | Prexasertib Cohort 4
Number analyzed (Participants) | 47 | 42 | 37 | 25
Months | 3.91 [3.68 to 5.68] | 3.71 [3.12 to 4.70] | 3.58 [1.87 to 3.91] | 3.71 [1.77 to 4.70]

7. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from the date of enrollment until death from any cause. If the participant is alive, lost to follow-up or withdrawn from study at the time of data analysis, OS data will be censored on the last date the participant is known to be alive.
Time Frame: Baseline to Date of Death from Any Cause (Up to 26 months)
Population: All randomized participants who received at least one dose of study drug and had overall survival data. Number of participants censored Cohort 1 = 18, Cohort 2 = 12, Cohort 3 = 12 and Cohort 4 = 4.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Prexasertib Cohort 1 | Prexasertib Cohort 2 | Prexasertib Cohort 3 | Prexasertib Cohort 4
Number analyzed (Participants) | 35 | 34 | 29 | 25
Months | 13.04 [7.46 to 19.25] | 14.32 [11.76 to 16.46] | 11.14 [7.23 to 16.43] | 8.18 [6.18 to 11.93]

ADVERSE EVENTS:
Time Frame: Baseline, upto 26 Months
Description: All randomized participants who received at least one dose.
Arm/Group | Prexasertib Cohort 1 | Prexasertib Cohort 2 | Prexasertib Cohort 3 | Prexasertib Cohort 4
All-Cause Mortality (participants affected / at risk) | 2/53 | 1/46 | 1/41 | 1/29
Serious Adverse Events (participants affected / at risk) | 23/53 | 17/46 | 19/41 | 15/29
Other Adverse Events (participants affected / at risk) | 53/53 | 44/46 | 39/41 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prexasertib Cohort 1 (N=53) | Prexasertib Cohort 2 (N=46) | Prexasertib Cohort 3 (N=41) | Prexasertib Cohort 4 (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 3 (4) | 5 (5) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 4 (4) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 4 (4) | 1 (1) | 3 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstruction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 5 (5) | 1 (1) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (2) | 2 (2) | 2 (3)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (11) | 0 (0) | 1 (6) | 1 (1)
Platelet count decreased (Investigations) | 1 (6) | 0 (0) | 1 (2) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (4) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prexasertib Cohort 1 (N=53) | Prexasertib Cohort 2 (N=46) | Prexasertib Cohort 3 (N=41) | Prexasertib Cohort 4 (N=29)
Anaemia (Blood and lymphatic system disorders) | 20 (64) | 17 (38) | 15 (40) | 12 (26)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 4 (7) | 1 (2) | 6 (10) | 4 (7)
Neutropenia (Blood and lymphatic system disorders) | 19 (40) | 10 (26) | 11 (24) | 10 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (83) | 14 (36) | 14 (34) | 7 (18)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 2 (3) | 0 (0) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2) | 5 (7)
Abdominal pain (Gastrointestinal disorders) | 14 (18) | 18 (40) | 11 (15) | 10 (14)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 2 (4) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 4 (6) | 2 (2) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1) | 5 (11) | 2 (3) | 2 (3)
Constipation (Gastrointestinal disorders) | 13 (19) | 12 (15) | 8 (13) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 19 (57) | 15 (19) | 7 (11) | 8 (20)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (4) | 4 (4) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 3 (5) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (54) | 24 (56) | 15 (33) | 16 (25)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (4) | 2 (2) | 1 (2) | 4 (5)
Vomiting (Gastrointestinal disorders) | 21 (29) | 13 (20) | 11 (36) | 14 (25)
Asthenia (General disorders) | 8 (19) | 8 (16) | 10 (38) | 4 (13)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 21 (84) | 19 (37) | 12 (17) | 12 (20)
Mucosal inflammation (General disorders) | 5 (8) | 1 (1) | 3 (5) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 3 (6) | 1 (1)
Oedema peripheral (General disorders) | 4 (5) | 3 (3) | 3 (3) | 1 (1)
Pain (General disorders) | 4 (4) | 2 (3) | 5 (6) | 3 (3)
Pyrexia (General disorders) | 13 (17) | 5 (6) | 7 (16) | 8 (9)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (9) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (9) | 3 (5) | 0 (0) | 4 (4)
Viral infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (5) | 6 (9) | 4 (5) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 3 (4) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 3 (3) | 1 (1) | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 3 (4) | 2 (2) | 3 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (11) | 9 (13) | 5 (9) | 1 (1)
Platelet count decreased (Investigations) | 8 (37) | 7 (17) | 7 (28) | 3 (4)
Weight decreased (Investigations) | 2 (2) | 3 (4) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 3 (7) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 12 (14) | 12 (21) | 9 (12) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (11) | 5 (10) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (12) | 2 (4) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6) | 3 (3) | 3 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (11) | 5 (6) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 8 (14) | 6 (7) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 3 (4) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (13) | 2 (2) | 2 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (4) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 5 (8) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 8 (9) | 10 (21) | 3 (7) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2) | 4 (4)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 3 (5) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 2 (2) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 7 (8) | 4 (5) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (9) | 6 (7) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 1 (4) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 2 (2) | 3 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT03414047/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT03414047/SAP_001.pdf